CLINICAL TRIAL: NCT07301775
Title: A Randomised Controlled Trial Comparing Efficacy of Single Versus Multiple Intravitreal Anti-VEGF Injections to Prevent Diabetic Retinopathy Progression in Patients Undergoing Cataract Surgery
Brief Title: Comparing Single Versus Multiple Anti-VEGF Injections in Diabetic Patients Undergoing Cataract Surgery
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Ahmad Zeeshan Jamil (Other)
Collaborators: Sahiwal medical college sahiwal (Other Government)
Responsible Party: Sponsor-Investigator, Ahmad Zeeshan Jamil, Professor and Head, Department of Ophthalmology, University of Health Sciences Lahore
Organization: University of Health Sciences Lahore (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 290/IRB/SLMC/SWL
Record Dates: First submitted 2025-12-10; First posted 2025-12-24 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Diabetic Retinopathy (DR); Diabetic Macular Edema (DME); Cataract; Phacoemulfisication+IOL Implantation; Intravitreal Injection
Keywords: Vascular endothelial growth factor; Aflibercept; Cataract Extraction; Intravitreal Injection; Phacoemulsification; Diabetic retinopathy; Diabetic macular edema; Intraocular lens implantation
MeSH Terms: conditions — Diabetic Retinopathy; Cataract | interventions — aflibercept

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Single injection Group (Active Comparator): Intravitreal Aflibercept 2mg/0.05ml injection will be given by standard technique at the end of Phacoemulsification with Intraocular lens implantation
  Interventions: Drug: Aflibercept (Eylea)
- Multiple Injection Group (Experimental): This group will receive Aflibercept intravitreal injection 2mg/0.05ml by standard technique at the end of the phacoemulsification with intraocular lens implantation and then at 1st, and 2nd months postoperatively.
  Interventions: Drug: Aflibercept (Eylea)

INTERVENTIONS:
Drug: Aflibercept (Eylea) — Single injection group will receive aflibercept intravitreal injection 2mg/0.05ml by the standard technique at the end of phacoemulsification with intraocular lens implantation. Multiple injection group will receive aflibercept intravitreal injection 2mg/0.05ml by standard technique at the end of phacoemulsification with intraocular lens implantation and then at 1st, and 2ndmonths postoperatively.

SUMMARY:
Objective of this randomised controlled trial is to compare the efficacy of a single per operative anti VEGF injection with repeated postoperative anti VEGF injections in the prevention of diabetic retinopathy progression after cataract surgery.

This Randomised Controlled Trial (RCT) will be conducted at Sahiwal Teaching Hospital and University College of Medicine & Dentistry Lahore. Duration of study will be from January 2026 to September 2026. This study will be single blind and parallel group research.

The study will include diabetic patients of both sexes ≥ 40 years of age presenting with non-proliferative diabetic retinopathy and cataract.

Exclusion criteria include proliferative diabetic retinopathy, center-involving diabetic macular oedema (DME), poor glycemic control (HbA1c >9%), glaucoma, uveitis, prior ocular surgery or laser, and recent systemic thromboembolic events.

Subjects will be randomly divided into two groups, each containing 83 subjects. Standard phacoemulsification with intraocular lens implantation will be performed in all participants.

A single intra vitreal Aflibercept injection ( 2mg/0.05 ml ), will be given to group 1 participants. While, group 2 participants will receive an intra operative injection plus two additional injections at 1 month and 2 months postoperatively.

For all participants, follow up will be performed at 1 week, 1 month, 2 month, 3 month and 6 month.

Primary Outcome include progression of diabetic retinopathy (DR) severity (≥1 stage according to the guidelines of the international clinical diabetic retinopathy disease severity scale ICDR) or onset/progression of DME.

Secondary Outcomes include changes in best corrected visual acuity, changes in central macular thickness (CMT), and need for rescue treatment.

SPSS version 26 will be utilised to analyse the data. P ≤ 0.05 will be taken as statistically significant. Qualitative variable like diabetic retinopathy grading and diabetic macular oedema status will be analysed by utilising Pearson's chi-square test. Quantitative variables like central macular thickness will be analysed by employing t-test.

DETAILED DESCRIPTION:
Title A randomized controlled trial comparing efficacy of single versus multiple intravitreal anti VEGF injections to prevent diabetic retinopathy progression in patients undergoing cataract surgery

Brief Title Comparing single versus multiple anti VEGF injections in diabetic patients undergoing cataract surgery.

Topic of interest: Role of anti VEGF injections in preventing progression of diabetic retinopathy in patients undergoing cataract surgery.

Research gap: A comparison of different dosing protocols in preventing progression of diabetic retinopathy in patients undergoing cataract surgery is not available.

Research question Among patients with diabetic retinopathy undergoing cataract surgery, does a single intravitreal anti-VEGF injection or a multiple-injection protocol more effectively prevent disease progression? Introduction Diabetic retinopathy is an emerging leading cause of defective vision worldwide . Systemic risk factors are important in causation of diabetes related visual morbidity . Cataract surgery is the most commonly performed elective surgery world-wide . Cataract surgery leads to increase in inflammatory mediators including vascular endothelial growth factor (VEGF) that can lead to progression of diabetic retinopathy . Before planning cataract surgery, diabetic control is utmost important . Despite good glycaemic control cataract surgery can result in progression of diabetic retinopathy and leading to unsatisfactory visual outcomes despite good cataract surgery . Different measures are taken to suppress inflammation associated with cataract surgery. Phacoemulsification in contrast to extracapsular cataract surgery leads to less inflammation and early recovery. Use of perioperative and postoperative steroids and nonsteroidal anti-inflammatory drugs significantly result in less post cataract surgery inflammation and hence less chances of progression of diabetic retinopathy . Despite all these measures diabetic retinopathy does show progression after cataract surgery . It has been shown that per operative use of anti VEGF injection prevents the progression of diabetic retinopathy. Anti-VEGF agents stop the action of VEGF by binding to the VEGF chemical, thereby preventing it from attaching to its receptors . But action of anti VEGF injections is short lived. It has been shown that post operative inflammation can persist many weeks after cataract surgery especially in diabetic patients. So there should be a need of repeated anti VEGF injection to completely mitigate the effects of cataract surgery induced inflammation in the progression of diabetic retinopathy . Currently there is no consensus on dosing protocol of anti-VEGF agents.

One study demonstrated that after cataract surgery 30.6% cases showed progression in diabetic retinopathy . In another study 38.2% eyes showed progression in diabetic retinopathy six months after cataract surgery .

According to our hypothesis, repeated postoperative anti VEGF injections prevent diabetic retinopathy progression to a greater extent than a single per operative anti-VEGF injection.

Objective of this randomized controlled trial is to compare the efficacy of a single per operative anti VEGF injection with repeated postoperative anti VEGF injections in the prevention of diabetic retinopathy progression after cataract surgery.

Methodology This randomized controlled trial will be conducted at the Sahiwal Teaching Hospital, Sahiwal and University College of Medicine & Dentistry Lahore from January 2026 to September 2026. The study will follow the guidelines of the Declaration of Helsinki. The study protocol will be approved by institutional review boards of respective hospitals. Written informed consent will be taken from all the subjects. The first subject will be recruited in January 2026, and the last subject will be recruited in June 2026. Three more months will be required to complete the final follow-up of the last subject.

The study will include diabetic patients of both sexes ≥ 40 years of age presenting with non-proliferative diabetic retinopathy and cataract.

Exclusion criteria will include the presence of proliferative diabetic retinopathy (PDR), diabetic macular oedema involving foveal centre, history of intraocular surgery or laser photocoagulation or prior anti-VEGF injection therapy in the study eye within past six months, history of intraocular inflammation (uveitis), glaucoma, mature cataract preventing satisfactory fundus examination preoperatively, poor glycaemic control (HbA1c>9%), pregnant and lactating women, known allergy to aflibercept (anti-VEGF used) and systemic thromboembolic events (stroke, myocardial infarction) within the last three months.

A comprehensive history will be obtained, including patient's presenting complaints, prior treatment history and risk factors associated with diabetic retinopathy.

Comprehensive ocular examination, including visual acuity by Snellen's chart, intraocular pressure by Goldmannn tonometer, and examination of the anterior and posterior segments, will be performed. Preoperative macular OCT scan will be performed with HOCT-1/1F(Huvitz). Grading of diabetic retinopathy will be done according to the guidelines of the international clinical diabetic retinopathy disease severity scale (ICDR) .

The sample size is calculated to detect a statistically significant difference in the progression of diabetic retinopathy between the two study groups. The calculation is based on the results of a pilot study conducted prior to the full-scale research.

Seventy-five participants will be included in each group. To account for a potential dropout/attrition rate of 10%, the final sample size is adjusted to include 83 patients in each group. Therefore, the study requires a total of 166 patients (83 patients per group) to achieve 80% power at a 5% significance level.

Randomization will be performed by employing a sequentially numbered, opaque, sealed envelope technique. Patients will be divided into two groups with 83 subjects in each group. Both groups will undergo standard phacoemulsification with intraocular lens implantation. Group 1 will receive aflibercept intravitreal injection 2mg/0.05ml by the standard technique at the end of the procedure. Group 2 will receive aflibercept intravitreal injection 2mg/0.05ml by standard technique at the end of the procedure and then at 1st, and 2ndmonths postoperatively.

This will be a single blind, parallel group, randomized controlled trial with 1:1 allocation, in which the outcome assessors will be unaware of the intervention.

Standard phacoemulsification with intraocular lens implantation will be performed by two surgeons, one surgeon at Sahiwal Teaching Hospital Sahiwal and other surgeon at University College of Medicine & Dentistry Lahore. A combination of steroid and antibiotic eye drops will be administered eight times per day during the first postoperative week. The dosing will be tapered off during the next three weeks.

Follow-up will be performed at one week, one month, two months, three months and six months postoperatively. The progression of diabetic retinopathy, status of diabetic macular oedema centre involving, best corrected visual acuity, centre macular thickness will be recorded. The posterior segment will be examined with the help of a super-field lens and oct will be performed at each visit.

The primary outcomes include the change in diabetic retinopathy severity ≥1 stage increase in ICDR scale or onset or progression of diabetic macular oedema. Secondary outcomes include changes in best corrected visual acuity, changes in central macular thickness and need for rescue treatment that is development of proliferative diabetic retinopathy and centre involving macular oedema causing decline in best corrected visual acuity (BCVA). Rescue treatment will include anti-VEGF injections and retinal laser photocoagulation. Centre involving macular oedema is defined as central 1 mm subfield thickness more that 300 microns. All patients will be followed up for six months or until the study participant will need rescue treatment in case of development of high-risk PDR or centre involving diabetic macular oedema causing decline in BCVA.

All information will be collected using a specially designed proforma and entered into SPSS version 26. Qualitative variables, such as sex, diabetic retinopathy grading, status of diabetic macular oedema, and final visual acuity, will be presented as frequencies and percentages. Quantitative variables, such as age and central macular thickness, will be presented as mean and standard deviation.

In this prospective study we shall investigate the differences in the changes in diabetic retinopathy and diabetic macular oedema between two distinct groups. Furthermore, we shall compare the change in visual acuity and the central macular thickness at the final follow-up visit between the two groups. For qualitative variables (frequency of eyes with different grades of diabetic retinopathy, Frequency of eyes with changes in macular oedema, and frequency of eyes with improved visual acuity), Pearson's chi-square test will be used to carry out the statistical analysis. For quantitative variables like central macular thickness t test will be used for statistical analysis. Statistical significance will be set at P ≤ 0.05.

ELIGIBILITY:
Inclusion Criteria:

* diabetic patients of both sexes ≥ 40 years of age presenting with non-proliferative diabetic retinopathy and cataract

Exclusion Criteria:

* presence of proliferative diabetic retinopathy (PDR), diabetic macular oedema involving foveal centre, history of intraocular surgery or laser photocoagulation or prior anti-VEGF injection therapy in the study eye within past six months, history of intraocular inflammation (uveitis), glaucoma, mature cataract preventing satisfactory fundus examination preoperatively, poor glycaemic control (HbA1c>9%), pregnant and lactating women, known allergy to aflibercept (anti-VEGF used) and systemic thromboembolic events (stroke, myocardial infarction) within the last three months.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 166 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Change from basseline in diabetic retinopathy severity at 6 months | Within six months after phacoemulsification with intraocular lens implantation
  Change in diabetic retinopathy severity ≥1 stage increase in international clinical diabetic retinopathy disease severity scale (ICDR) or onset or progression of diabetic macular oedema

CONTACTS AND LOCATIONS:
Overall Officials: AHMAD ZEESHAN JAMIL, FCPS, FRCS, FCPS(VRO), Principal Investigator — Sahiwal Medical College and Sahiwal Teaching Hospital Sahiwal
Locations (2):
- Pakistan (2):
  - University College of Medicine and Dentistry (UCMD), Lahore, Punjab Province
  - Sahiwal Medical College and Sahiwal Teaching Hospital, Sahiwal, Punjab, Pakistan

IPD SHARING:
Plan to Share IPD: Yes
Yes. De-identified individual participant data (IPD) underlying the main results (baseline characteristics, intervention details, and primary/secondary outcomes) will be made available upon reasonable request to the principal investigator after publication. Data will be shared through institutional repositories subject to IRB approval and data-sharing agreements.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: De-identified individual participant data (IPD) will be made available beginning 6 months after publication of the primary results and will remain accessible for a period of 2 years following study completion.
Access Criteria: De-identified individual participant data (IPD) and supporting documents (protocol, SAP, consent template) will be available to qualified researchers affiliated with academic or medical institutions. Access will be granted upon IRB approval and execution of a data-sharing agreement. Data will be shared via secure institutional repository within 6-12 months after publication and remain available for 2 years.
URL: https://eyecon.pk

REFERENCES:
- [Background] Wilkinson CP, Ferris FL 3rd, Klein RE, Lee PP, Agardh CD, Davis M, Dills D, Kampik A, Pararajasegaram R, Verdaguer JT; Global Diabetic Retinopathy Project Group. Proposed international clinical diabetic retinopathy and diabetic macular edema disease severity scales. Ophthalmology. 2003 Sep;110(9):1677-82. doi: 10.1016/S0161-6420(03)00475-5. PMID 13129861
- [Background] Pollack A, Dotan S, Oliver M. Progression of diabetic retinopathy after cataract extraction. Br J Ophthalmol. 1991 Sep;75(9):547-51. doi: 10.1136/bjo.75.9.547. PMID 1911658
- [Background] Chung J, Kim MY, Kim HS, Yoo JS, Lee YC. Effect of cataract surgery on the progression of diabetic retinopathy. J Cataract Refract Surg. 2002 Apr;28(4):626-30. doi: 10.1016/s0886-3350(01)01142-7. PMID 11955902
- [Background] Starr MR, Mahr MA, Smith WM, Iezzi R, Barkmeier AJ, Bakri SJ. Outcomes of Patients With Active Diabetic Macular Edema at the Time of Cataract Surgery Managed With Intravitreal Anti-Vascular Endothelial Growth Factor Injections. Am J Ophthalmol. 2021 Sep;229:194-199. doi: 10.1016/j.ajo.2021.04.002. Epub 2021 Apr 20. PMID 33852907
- [Background] Hu W, Ni L, Ying H, Zhang Z, Tu S, Tao Y, Chen L. Efficacy of fluocinolone acetonide implant in diabetic macular edema patients previously treated with dexamethasone implant: A systematic review and meta-analysis. Pak J Med Sci. 2025 Aug;41(8):2388-2398. doi: 10.12669/pjms.41.8.12675. PMID 40980399
- [Background] Cheema RA, Al-Mubarak MM, Amin YM, Cheema MA. Role of combined cataract surgery and intravitreal bevacizumab injection in preventing progression of diabetic retinopathy: prospective randomized study. J Cataract Refract Surg. 2009 Jan;35(1):18-25. doi: 10.1016/j.jcrs.2008.09.019. PMID 19101420
- [Background] Haddad JE, Sabbakh NA, Macaron MM, Shaaban H, Bourdakos NE, Shi A, Saad B, Nakanishi H, Than CA, Daoud YJ. NSAIDs and Corticosteroids for the Postoperative Management of Age-Related Cataract Surgery: A Systematic Review and Meta-analysis. Am J Ophthalmol. 2024 Apr;260:1-13. doi: 10.1016/j.ajo.2023.09.027. Epub 2023 Oct 4. PMID 37797866
- [Background] Kropp M, Golubnitschaja O, Mazurakova A, Koklesova L, Sargheini N, Vo TKS, de Clerck E, Polivka J Jr, Potuznik P, Polivka J, Stetkarova I, Kubatka P, Thumann G. Diabetic retinopathy as the leading cause of blindness and early predictor of cascading complications-risks and mitigation. EPMA J. 2023 Feb 13;14(1):21-42. doi: 10.1007/s13167-023-00314-8. eCollection 2023 Mar. PMID 36866156
- [Background] Kaur A, Kumar R, Sharma A. Diabetic Retinopathy Leading to Blindness- A Review. Curr Diabetes Rev. 2024;20(9):e240124225997. doi: 10.2174/0115733998274599231109034741. PMID 38275038
- [Background] Han X, Zhang J, Liu Z, Tan X, Jin G, He M, Luo L, Liu Y. Real-world visual outcomes of cataract surgery based on population-based studies: a systematic review. Br J Ophthalmol. 2023 Aug;107(8):1056-1065. doi: 10.1136/bjophthalmol-2021-320997. Epub 2022 Apr 11. PMID 35410876
- [Background] Lee SH, Tseng BY, Wu MC, Wang JH, Chiu CJ. Incidence and Progression of Diabetic Retinopathy After Cataract Surgery: A Systematic Review and Meta-Analysis. Am J Ophthalmol. 2025 Jan;269:105-115. doi: 10.1016/j.ajo.2024.08.017. Epub 2024 Aug 22. PMID 39179126
- [Background] Rachmilevich A, Yanculovich N, Hazan I, Tsumi E, Liberty IF. Glycemic control and macular edema in patients undergoing cataract surgery. Prim Care Diabetes. 2023 Feb;17(1):55-59. doi: 10.1016/j.pcd.2022.12.004. Epub 2023 Jan 2. PMID 36599797
- [Background] Sruthi R, Saikumar SJ, Gopalakrishnan M. Progression of diabetic retinopathy following uncomplicated phacoemulsification: A prospective study from South India. Oman J Ophthalmol. 2024 Feb 21;17(1):72-77. doi: 10.4103/ojo.ojo_292_22. eCollection 2024 Jan-Apr. PMID 38524349
- [Background] Wu J, Zhou Y, Zhen F, Wang S, Li Q, Dong S. Management after cataract surgery for patients with diabetic retinopathy: a systematic review and meta-analysis. Int Ophthalmol. 2024 Apr 1;44(1):166. doi: 10.1007/s10792-024-02981-6. PMID 38557801
- Available data/document: Individual Participant Data Set — http://www.eyecon.pk